CLINICAL TRIAL: NCT05086055
Title: Training the Surviving Neural Network to Create New Synaptic Connections That Can Maximize Restoration of Motor Functions After Stroke
Brief Title: Rehabilitation of Stroke Patients for Maximal Neurological Restoration
Acronym: PROTEQT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other); OsloMet (Unknown)
Responsible Party: Sponsor
Other Study IDs: 171264
Record Dates: First submitted 2021-05-25; First posted 2021-10-20 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Stroke
Keywords: Rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stroke patients: Stroke patients admitted to the stroke unit, St Olav´s hospital, Trondheim, Norway, without previous stroke, neurological disease or central nervous system (CNS) trauma, will be eligible for inclusion into the study. The planned cohort size is 135 patients.
  Interventions: Behavioral: Kinematic movement analysis
- healthy volunteers: Age and gender matched controls without previous CNS disease or trauma are eligible for inclusion into the study. Estimated cohort size is 45 individuals. Volunteers will be recruited through announcement in local newspaper.
  Interventions: Behavioral: Kinematic movement analysis

INTERVENTIONS:
Behavioral: Kinematic movement analysis — moving arm/leg while registration with electromyography, electroencephalogram, accelerometers, functional near infrared spectroscopy and 3 dimensional video registration of hand, arm, foot and leg movements.

SUMMARY:
Multimodal imaging of stroke patients. Patients included in the study will be investigated with multiparametric imaging tools including MRI and EEG imaging. Improvements in motor skills will be monitored clinically.

DETAILED DESCRIPTION:
We aim to (i) quantify the size of the brain lesion and assess the surviving functional neural network connections; (ii) Analyze the type and degree of inflammation initiated by the stroke-induced brain lesion. We will stratify inflammation according to lesion volume, surviving functional neural network connections, age, NIHSS and Modified Rankin Scale (mRS) and analyze how inflammation markers change during rehabilitation; (iii) Train the surviving neural network to create new synaptic connections that can maximize restoration of motor functions; (iv) Apply and develop advanced mathematical and computational methods to model and predict how stroke rehabilitation can rewire the neural network connections to best facilitate restoration of lost motor function.

ELIGIBILITY:
Inclusion Criteria:

* subcortical strokes resulting in arm motor deficits.
* admitted to the stroke unit, St Olav´s Hospital during 2021-2023

Exclusion Criteria:

* Previous stroke
* neurodegenerative disease
* brain tumors
* previous neurotrauma or brain operation
* aphasia
* cognitive dysfunction and claustrophobia preventing MRI examinations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18-years or older of both sexes with subcortical strokes resulting in arm motor deficit, admitted to the stroke unit, St Olav´s Hospital during 2020-2023. All patients admitted to the stroke unit will be scored according to National Institute of Health Score Scale (NIHSS) and the modified Rankin score (mRS) to establish the baseline clinical assessment of neurological dysfunction prior to inclusion
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-11-11 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Changes in brain volume | 6 months
  Stroke induced brain volume changes (mm3) will be measured using magnetic resonance imaging (MRI) at 1 day and 6 months post-stroke.
Stroke induced changes in brain activity. | 6 months
  Document longitudinal changes in brain activity using EEG. Changes will be measured in cycles/second (Hertz, Hz).
Changes in inflammatory activity in brain | 6 months
  Markers of post-stroke inflammation will be measured in pg/ml and ng/ml.
muscle function | 6 months
  Longitudinal kinematic profiling. Electromyography measurements of muscle function post-stroke will be measured in cycles/second (Hz) and amplitude (mm). Extension and flexion of arm will be measured in cm. Joint angles will be measured in degrees. Speed of flexion and extension will be measured in cm/second

CONTACTS AND LOCATIONS:
Overall Officials: Axel Sandvig, PhD prof, Principal Investigator — Norwegian University of Science and Technology; Jorunn Helbostad, PhD prof, Study Director — Norwegian University of Science and Technology; Bent Indredavik, PhD prof, Study Director — St. Olavs Hospital
Locations (3):
- Norway (3):
  - OsloMet, Oslo
  - NextMove, NTNU, Trondheim
  - St Olavs Hospital Stroke Unit, Trondheim

IPD SHARING:
Plan to Share IPD: No